CLINICAL TRIAL: NCT01680341
Title: A Trial Comparing the Efficacy and Safety of Two Different Titration Algorithms for Insulin Degludec/Insulin Aspart in Subjects With Type 2 Diabetes Mellitus Previously Treated With Insulin Glargine (BOOST®: SIMPLE vs. STEPWISE)
Brief Title: Comparison of the Efficacy and Safety of Two Different Dose Adjustment Regimens for Insulin Degludec/Insulin Aspart in Subjects With Type 2 Diabetes Mellitus Previously Treated With Insulin Glargine
Acronym: BOOST®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3941; 2012-000373-23 (EudraCT Number); U1111-1127-4114 (Other: WHO)
Record Dates: First submitted 2012-08-31; First posted 2012-09-07 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp Simple (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- IDegAsp Step wise (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Twice weekly self-titration at intervals of 3-4 days, based upon a single pre-breakfast and pre-dinner SMPG (self-measured plasma glucose) value. For subcutaneous (s.c., under the skin) administration.
  Other Names: IDegAsp
  Arms: IDegAsp Simple
Drug: insulin degludec/insulin aspart — Once weekly self-titration based upon the lowest of 3 pre-breakfast and 3 pre-dinner SMPG (self-measured plasma glucose) values. For subcutaneous (s.c., under the skin) administration.
  Other Names: IDegAsp
  Arms: IDegAsp Step wise

SUMMARY:
This trial is conducted in Africa, Asia, Europe and the United States of America (USA).

The aim of the trial is to compare the efficacy and safety of two different titration algorithms for insulin degludec/insulin aspart (IDeg/IAsp) in subjects with type 2 diabetes mellitus previously treated with insulin glargine.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed clinically) for at least 24 weeks prior to Visit 2 (randomisation)
* Currently treated with IGlar (Insulin Glargine) and up to 3 oral antidiabetic drugs (OADs) (metformin, DPP-4 inhibitor, sulphonylurea/glinide or alpha-glucosidase inhibitor). All antidiabetic treatments should have been ongoing for at least 12 weeks prior to Visit 2 (randomisation) and doses should have been stable in this period of time
* Glycosylated haemoglobin (HbA1c) 7.0-10.0% (both inclusive) by central laboratory analysis
* Body mass index (BMI) below or equal to 40 kg/m^2

Exclusion Criteria:

* Treatment with glucagon-like peptide 1 (GLP-1) receptor agonists or thiazolidinediones (TZDs) both within the last 12 weeks prior to Visit 2 (randomisation)
* Stroke; heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty; all within the last 24 weeks prior to Visit 2 (randomisation)
* Uncontrolled or untreated severe hypertension defined as systolic blood pressure above or equal to 180 mmHg and/or diastolic blood pressure above or equal to 100 mmHg
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during last 12 months) or hypoglycaemic unawareness as judged by the investigator
* Life-threatening disease (e.g. cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2012-08-31 (Actual); Primary Completion 2013-08-22 (Actual); Study Completion 2013-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (44):
- United States (27):
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Suwanee, Georgia
  - Novo Nordisk Investigational Site, Avon, Illinois
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Tacoma, Washington
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
- Algeria (3):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Tizi Ouzou
- Germany (6):
  - Novo Nordisk Investigational Site, Erdmannhausen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saint Ingbert
- Malaysia (3):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Kuala Selangor
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Denizli
  - Novo Nordisk Investigational Site, Gaziantep
  - Novo Nordisk Investigational Site, Hatay
  - Novo Nordisk Investigational Site, Istanbul

REFERENCES:
- [Result] Bode BW, Buse JB, Fisher M, Garg SK, Marre M, Merker L, Renard E, Russell-Jones DL, Hansen CT, Rana A, Heller SR; BEGIN(R) Basal-Bolus Type 1 trial investigators. Insulin degludec improves glycaemic control with lower nocturnal hypoglycaemia risk than insulin glargine in basal-bolus treatment with mealtime insulin aspart in Type 1 diabetes (BEGIN((R)) Basal-Bolus Type 1): 2-year results of a randomized clinical trial. Diabet Med. 2013 Nov;30(11):1293-7. doi: 10.1111/dme.12243. Epub 2013 Jun 17. PMID 23710902
- [Result] Haluzik M, Fulcher G, Pieber TR, Bardtrum L, Tutkunkardas D, Rodbard HW. The co-formulation of insulin degludec and insulin aspart lowers fasting plasma glucose and rates of confirmed and nocturnal hypoglycaemia, independent of baseline glycated haemoglobin levels, disease duration or body mass index: A pooled meta-analysis of phase III studies in patients with type 2 diabetes. Diabetes Obes Metab. 2018 Jul;20(7):1585-1592. doi: 10.1111/dom.13261. Epub 2018 Mar 25. PMID 29451706
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- [Derived] Gerety G, Bebakar WM, Chaykin L, Ozkaya M, Macura S, Herslov ML, Behnke T. TREATMENT INTENSIFICATION WITH INSULIN DEGLUDEC/INSULIN ASPART TWICE DAILY: RANDOMIZED STUDY TO COMPARE SIMPLE AND STEP-WISE TITRATION ALGORITHMS. Endocr Pract. 2016 May;22(5):546-54. doi: 10.4158/EP15893.OR. Epub 2015 Dec 31. PMID 26720250
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 43 sites in 5 countries: Algeria (3 sites), Germany (5 sites), Malaysia (3 sites), Turkey (3 sites), and United States (29 sites).
Pre-assignment Details: While entering the treatment period the subjects discontinued insulin glargine (IGlar) and sulfonylurea (SU)/glinides (if administered) but continued treatment with up to 3 other oral antidiabetic drugs (OADs) as prescribed.
Groups:
- IDegAsp Simple: Insulin degludec/insulin aspart (IDegAsp) was injected subcutaneously (s.c.) in either abdomen, upper arm (deltoid area) or thigh. A pre-filled pen injector (PDS290) was used to administer IDegAsp. During treatment period subjects were allowed to continue up to 3 (oral antidiabetic drugs) OADs, except insulin glargine, sulphonylurea and glinides. In the IDegAsp twice daily (BID) simple titration algorithm arm, self-titration was performed twice weekly at intervals of 3-4 days and based upon a single pre-breakfast and pre-dinner self-measured plasma glucose (SMPG) value.
- IDegAsp Step Wise: IDegAsp was injected subcutaneously (s.c.) in either abdomen, upper arm (deltoid area) or thigh. A pre-filled pen injector (PDS290) was used to administer IDegAsp. During treatment period subjects were allowed to continue up to 3 (oral antidiabetic drugs) OADs, except insulin glargine, sulphonylurea and glinides. In the IDegAsp twice daily (BID) stepwise titration algorithm arm, self-titration was done once weekly based on the lowest of 3 pre-breakfast and 3 pre-dinner SMPG values (measurements on 3 consecutive days prior to titration).
Period: Overall Study
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Started | 136 | 136
Exposed | 135 (One (1) subject withdrew consent prior to exposure to trial product.) | 134 (Two (2) subjects withdrew consent prior to exposure to trial product.)
Completed | 115 | 119
Not Completed | 21 | 17
Not completed — Adverse Event | 3 | 2
Not completed — Unclassified | 18 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp Simple | IDegAsp Step Wise | Total
Number analyzed (Participants) | 136 | 136 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (9.8) | 59.1 (9.4) | 58.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 53 | 113
  Male | 76 | 83 | 159
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.2 (0.9) | 8.2 (0.9) | 8.2 (0.9)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 7.8 (2.3) | 8.1 (3.0) | 8.0 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin) (%)
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects. Missing data were imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Percent (%) glycosylated haemoglobin
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 136 | 136
Percent (%) glycosylated haemoglobin | -1.45 (0.09) | -1.33 (0.09)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline in fasting plasma glucose (FPG) after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects. Missing data were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 136 | 136
mmol/L | -1.68 (0.23) | -1.98 (0.23)

3. Secondary Outcome: Subjects With HbA1c Below 7.0%
Description: Number of subjects with HbA1c below 7% after 26 weeks of treatment.
Time Frame: Week 26
Population: The full analysis set (FAS) included all randomised subjects. Missing data were imputed using LOCF.
Measure: Number; unit: Subjects
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 136 | 136
Subjects | 91 | 85

4. Secondary Outcome: Percentage of Subjects With HbA1c Below 7.0% Without Confirmed Hypoglycaemia
Description: Percentage of subjects with HbA1c below 7% without confirmed hypoglycaemic episodes after 26 weeks of treatment.
Time Frame: Week 26
Population: The full analysis set (FAS) included all randomised subjects. Missing data were imputed using LOCF. Twenty five (25) subjects did not contribute to statistical analysis as Endpoint was only defined for subjects exposed for at least 12 treatment weeks.
Measure: Number; unit: percentage of subjects
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 122 | 125
percentage of subjects | 25.4 | 32.0

5. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: A Treatment Emergent Adverse Event (TEAE) was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Time Frame: Weeks 0-28
Population: The safety analysis set included all subjects who received at least one dose of the investigational product.
Measure: Number; unit: number of events
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 135 | 134
number of events | 242 | 286

6. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes
Description: Confirmed hypoglycaemic episodes consisted of episodes of severe hypoglycaemia and minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Weeks 0-27
Population: The safety analysis set included all subjects who received at least one dose of the investigational product.
Measure: Number; unit: episodes
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 135 | 134
episodes | 552 | 323

7. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes in the Maintenance Period
Description: Confirmed hypoglycaemic episodes in the maintenance period (from Week 16 to the end of the trial including follow-up [Week 27]) consisted of episodes of severe hypoglycaemia and minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: From week 16 to end of trial including follow-up (week 27)
Population: The safety analysis set included all subjects who received at least one dose of the investigational product. Subjects in maintenance period were included in this analysis.
Measure: Number; unit: episodes
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 121 | 124
episodes | 230 | 143

8. Secondary Outcome: Number of Treatment Emergent Nocturnal (00:01-05:59) Confirmed Hypoglycaemic Episodes
Description: Confirmed hypoglycaemic episodes consisted of episodes of severe hypoglycaemia and minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes were defined as occurring between 00:01 and 05:59 am.
Time Frame: Weeks 0-27
Population: The safety analysis set included all subjects who received at least one dose of the investigational product.
Measure: Number; unit: episodes
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Number analyzed (Participants) | 135 | 134
episodes | 82 | 49

ADVERSE EVENTS:
Time Frame: The adverse events were collected from week 0 to Week 28.
Description: The safety analysis set included all subjects who received at least one dose of the investigational product.
Arm/Group | IDegAsp Simple | IDegAsp Step Wise
Serious Adverse Events (participants affected / at risk) | 7/135 | 10/134
Other Adverse Events (participants affected / at risk) | 45/135 | 53/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp Simple (N=135) | IDegAsp Step Wise (N=134)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp Simple (N=135) | IDegAsp Step Wise (N=134)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 8 (12)
Bronchitis (Infections and infestations) | 6 (6) | 7 (7)
Influenza (Infections and infestations) | 5 (5) | 12 (12)
Nasopharyngitis (Infections and infestations) | 12 (16) | 20 (23)
Upper respiratory tract infection (Infections and infestations) | 14 (16) | 10 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (9)
Headache (Nervous system disorders) | 9 (10) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.